CLINICAL TRIAL: NCT05876975
Title: Vaginal Axis on MRI After Laparoscopic Pectopexy Surgery: a Controlled Study
Brief Title: Vaginal Axis on Magnetic Resonance Imaging After Laparoscopic Pectopexy Surgery: a Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, fatih sahin, MD / Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 77
Record Dates: First submitted 2023-05-11; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Pelvic Organ Prolapse
Keywords: Magnetic resonance imaging (MRI); vaginal angle; vaginal axis; pelvic organ prolapse (POP)
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- procedure: laparoscopic pectopexy (Active Comparator): MRI evaluation will be conducted on eleven participants who underwent laparoscopic pectopexy surgery after one month.
  Interventions: Procedure: laparoscopic pectopexy
- Nulliparous women with no uterovaginal prolapsed (No Intervention): Ten nulliparous participants with no uterovaginal prolapsed will be evaluate by MRI

INTERVENTIONS:
Procedure: laparoscopic pectopexy — Women with pelvic organ prolapse and suitable indications underwent laparoscopic pectopexy.
  Arms: procedure: laparoscopic pectopexy

SUMMARY:
Pelvic organ prolapse (POP) is a major public health concern that adversely affects the physical and psychological well-being of women. In fact, the lifetime risk of POP surgery is 12.6%, highlighting the magnitude of the problem. The most common form of POP involves defects in the anterior vaginal wall accompanied by apical prolapse. The primary objective of surgical treatment for POP is to mitigate symptoms and restore the pelvic support anatomy. Normally, the vaginal axis is directed posteriorly towards the S3 and S4 vertebrae, lying relatively horizontally to the levator plate, and forming an angle of about 130º between the middle and lower vagina. Although sacrocolpopexy (SCP) is considered the gold standard for treating POP, it alters the normal anatomical position of the vaginal axis towards the sacral promontory, which may increase the abdominal pressure load on the anterior wall and cause urge symptoms or de novo anterior compartment prolapse. Similarly, sacrospinous ligament fixation (SSLF) increases the risk of anterior vaginal wall prolapse, as it deviates the vaginal axis towards the posterior. However, laparoscopic lateral mesh suspension has recently become popular because it preserves the normal position of the vaginal axis, preventing such complications. A previous study found that the pectineal ligament (Cooper's ligament) is composed of stronger and more durable tissue than the sacrospinous ligament and arcus tendineus of the fascia pelvis. This structure is robust and can hold sutures well, and it is possible to find sufficient material for a suture in the lateral part of the iliopectineal ligament, facilitating pelvic floor reconstruction. This segment of the ligament is located at the second sacral vertebra (S2) level, which is the optimal level for the physiological axis of the vagina. S2 level serves as the anchor point for the physiological axis of the vagina. Further studies have demonstrated that laparoscopic pectopexy provides outcomes comparable to those of laparoscopic sacrocolpopexy for supporting the apical compartment during intermediate follow-up duration. The current study aimed to investigate the level of anatomical correction following laparoscopic pectopexy and compare the vaginal axis of patients with apical genital prolapse to that of nulliparous women using magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a significant health concern that has a negative impact on the physical and psychological well-being of women. In fact, the lifetime risk of undergoing POP surgery is 12.6%. The most common form of POP involves defects in the anterior vaginal wall accompanied by apical prolapse. The primary goal of surgical treatment for POP is to alleviate symptoms and restore the anatomy of the pelvic support. The normal position of the vaginal axis is directed posteriorly towards the S3 and S4 vertebrae, lying relatively horizontally to the levator plate, and forming an angle of about 130º between the middle and lower vagina. Sacrocolpopexy (SCP) is considered the gold standard for treating POP, but it alters the normal anatomical position of the vaginal axis towards the sacral promontory, which may increase the abdominal pressure load on the anterior wall and cause urge symptoms or de novo anterior compartment prolapse. Although sacrospinous ligament fixation (SSLF) has promising long-term outcomes for correcting the apical anatomy, it increases the risk of anterior vaginal wall prolapse, like SCP, due to the deviation of the vaginal axis towards the posterior. Recently, laparoscopic lateral mesh suspension, which keeps the vaginal axis close to normal, has become popular. In a previous study, it was found that the pectineal ligament (Cooper's ligament) is composed of stronger and more durable tissue than the sacrospinous ligament and arcus tendineus of the fascia pelvis. This structure is robust and can hold sutures well. Sufficient material for a suture can also be found in the lateral part of the iliopectineal ligament, making pelvic floor reconstruction easier. This segment of the ligament is located at the second sacral vertebra (S2) level, which is the optimal level for the physiological axis of the vagina. S2 level is the anchor point for the physiological axis of the vagina. Further studies have demonstrated comparable outcomes for supporting the apical compartment at intermediate follow-up duration compared to laparoscopic sacrocolpopexy. This study aimed to investigate the level of anatomical correction following Laparoscopic pectopexy and compare the vaginal axis of patients with apical genital prolapse to that of nulliparous women using magnetic resonance imaging (MRI).

ELIGIBILITY:
In Intervention Group

Inclusion Criteria:

* Women diagnosed with apical pelvic organ prolapse (POP), who did not require an additional posterior colporrhaphy procedure, and desired to undergo uterus-preserving surgery were scheduled for laparoscopic pectopexy.

Exclusion Criteria:

* Women with uterine size greater than 10 cm or a pelvic mass that may alter or interfere with accurate measurement.
* Women with any congenital or acquired anatomical or reproductive anomaly.
* Women diagnosed with enterocele through transperineal ultrasound prior to enrollment.
* Women who require hysterectomy or concomitant pelvic organ prolapse (POP) or anti- incontinence procedure.
* Women with abnormal uterine bleeding.
* Women with abnormal cervical screening test results.

In Control Group

Inclusion Criteria:

* Nulliparous women without pelvic organ prolapse (asymptomatic grade 1 or less) who presented to the outpatient clinic with complaints other than POP symptoms (e.g., menstrual irregularity) were randomly selected and assigned as the control group.

Exclusion Criteria:

* Women who have given birth previously.
* Women with a history of pelvic organ prolapse or any pelvic floor disorders.
* Women who have undergone pelvic surgery.
* Women with any congenital or acquired anatomical or reproductive anomaly.
* Women with abnormal uterine bleeding.
* Women with abnormal cervical screening test results.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-06-04 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Anatomic Success | 3 months
  anatomic success will be evaluated by using magnetic resonance imaging. Vaginal axis (distance to spin ischiadic a and sacrum) will be measure on three plane

SECONDARY OUTCOMES:
Urge Symptoms stres incontinence | 3 month
  UDI-6 Th e UDI-6 was developed to evaluate the functions of the bladder and to establish which symptom causes the problem. It comprises 6 questions. Th e fi rst 2 questions are related to irritative symptoms (urgency, frequency, and pain), questions 3 and 4 are related to stress incontinence, and the last 2 questions are related to obstructive or voiding diffi culty symptoms. High UDI-6 scores show the severity of the urogenital complaints
Sexual functions | 3 month
  The FSFI evaluates sexual functioning in women and comprises of 19 questions with different answer choice scales referring the sexual life in the previous 4 weeks. The answer choices in the FSFI carry a number of points and are summed to obtain six domain scores and an overall score. For the latter, there is a threshold at 26.55 which means tFhat all values below are classed as indicating female sexual dysfunction (FSD). The domain scores are obtained as the sum of points attributed to questions in that domain multiplied by the domain factor.

CONTACTS AND LOCATIONS:
Overall Officials: fatih şahin, MD, Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang H, Shen J, Li S, Gao Z, Ke K, Gu P. The feasibility of uterine-vaginal axis MRI-based as evaluation of surgical efficacy in women with pelvic organ prolapse. Ann Transl Med. 2022 Apr;10(8):447. doi: 10.21037/atm-22-1173. PMID 35571410